CLINICAL TRIAL: NCT00704821
Title: A Phase 1b Study to Assess the Safety Profile, Pharmacokinetics, and Anti-VEGF Activity of PTC299 in Patients With Advanced Cancer
Brief Title: PTC299 for Treatment of Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTC299-ONC-004-AST
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: Advanced Cancer
Keywords: Cancer; PTC299; VEGF; Angiogenesis; Post-transcriptional control; Docetaxel
MeSH Terms: conditions — Neoplasms | interventions — emvododstat; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stage 1 (Experimental): In Stage 1, PTC299 will be given orally twice a day (BID) each day at about the same time each day for the first 28 days of each cycle. Each cycle will constitute a 4-week (28 days) period followed by a ≥2-week (14-day) washout period. Participants will be assigned to 0.3 milligrams (mg)/kilograms (kg)/dose BID, 0.6 mg/kg/dose BID, or 1.2 mg/kg/dose BID sequentially based on safety evaluations by the Sponsor's medical monitor in Cycle 1. Treatment cycles can continue if therapy appears to be safely offering tumor control to participant.
  Interventions: Drug: PTC299
- Stage 2 (Experimental): In Stage 2, PTC299 will be given BID or 3 times a day (TID) orally each day at about the same time each day; therefore, 84 (for BID) or 126 (for TID) doses of PTC299 will be delivered during the 6-week (42-day) period in each cycle. Each participant will be assigned to 100 mg/dose BID, 100 mg/dose TID, 120 mg/dose TID, 160 mg/dose TID, or 200 mg/dose TID sequentially based on safety evaluations by the Sponsor's medical monitor in Cycle 1. Treatment cycles can continue if therapy appears to be safely offering tumor control to participant.
  Interventions: Drug: PTC299
- Stage 3 (Experimental): In Stage 3, PTC299 will be given BID or TID (for total of 42 [for BID] or 63 [for TID] doses) orally about same time per day starting on Day 1 in each 3-week (21-day) cycle. Starting dose will be 1 dose level below maximum tolerated dose (MTD) from Stage 2 or 80 mg/dose BID if 100 mg/dose TID in Stage 2 exceeds MTD. Dose escalation will be based on safety evaluations by Sponsor's medical monitor in Cycle 1. Treatment cycles can continue if therapy appears to be safely offering tumor control to participant. Participants will also receive docetaxel as a 1-hour IV infusion on Day 1 per cycle at starting dose of 75 mg/m^2 with body surface area calculation based on body weight. Dose will be sequentially reduced to 60 and 50 mg/m^2 in participants with a docetaxel-related dose-limiting toxicity (DLT). Participants will be medicated with oral corticosteroids with docetaxel administration. Recommended dose is 8 mg BID dexamethasone for 3 days starting 1 day prior to docetaxel administration.
  Interventions: Drug: PTC299; Drug: Docetaxel
- Stage 4 (Experimental): In Stage 4, PTC299 will be given orally each day continuously starting on first day of each cycle at about same time per day; so, 42 doses of PTC299 will be delivered for 3 weeks (21-day) in Cycle 1 (BID dosing), and 84 doses will be delivered for 3-weeks (21-day) in Cycle 2 and beyond (TID dosing). For Cycle 1, participants will be assigned to 600, 800, or 1000 mg/dose BID sequentially based on safety evaluations by Sponsor's medical monitor at enrollment. For Cycle 2 and beyond, participants will receive PTC299 160 mg/dose TID. During Cycle 1, Cohort 1 participants will eat a meal containing of ≤15 grams (g) of dietary fat and Cohort 2 participants will eat a meal containing of ≤25 g of dietary fat prior to each dose of PTC299. If ≤2 of 6 participants had experienced DLT during Cycle 1 in either diet plan, then the dose will be escalated to 800 mg BID in Cohort 3 at the optimal diet. Treatment cycles can continue if therapy appears to be safely offering tumor control to participant.
  Interventions: Drug: PTC299

INTERVENTIONS:
Drug: PTC299 — Oral
Drug: Docetaxel — Intravenous infusion
  Arms: Stage 3

SUMMARY:
Formation of new blood vessels (angiogenesis) is important for tumor growth in advanced cancer. It is known that tumors make a protein called vascular endothelial growth factor (VEGF). VEGF stimulates the formation of blood vessels that supply the tumor with nutrients and oxygen. PTC299 is an oral investigational new drug that has been shown to decrease production of VEGF in animal models of human cancer. In these animal models, oral PTC299 administration decreases VEGF levels in the tumor and in the bloodstream, decreases blood vessel numbers in the tumor, and significantly slows or halts tumor growth. When given in combination with the chemotherapeutic drug, docetaxel, PTC299 increases the antitumor activity over use of docetaxel alone. Safety studies in research animals indicate good tolerability at doses and drug levels that are higher than those planned for the clinical studies. Results from Phase 1a studies in healthy volunteers indicate that PTC299 achieves levels of PTC299 in the bloodstream that are known to be active in animal models of human cancer. This Phase 1b study is designed to test the hypothesis that PTC299 will be tolerable and will show evidence of anti-VEGF and antitumor activity when administered orally to participants with cancer.

DETAILED DESCRIPTION:
The study will be conducted in 3 stages. In Stage 1 of the study, successive groups of 3 to 6 participants will receive progressively higher PTC299 dose levels; in this stage, treatment will be given in repeated 6-week cycles consisting of 4 weeks of oral PTC299 twice per day followed by a 2-week, no-drug period. In Stage 2, additional groups of 3 to 6 participants will be enrolled at tolerable dose levels to receive treatment in repeated 6-week cycles consisting of oral PTC299 administered 2 or 3 times per day continuously (that is, without the 2-week no-drug period as in Stage 1). In Stage 3, additional groups of 3 to 6 participants will be enrolled at tolerable dose levels to receive treatment in repeated 3-week cycles consisting of oral PTC299 administered 2 or 3 times per day continuously in combination with docetaxel (75 milligrams/meter squared [mg/m^2] intravenously [IV] every 3 weeks). All planned dose levels in all stages are expected to achieve circulating blood levels of PTC299 known to be active in animal models of human cancer. Treatment for each participant can continue as long as the therapy appears to be safely offering tumor control to that participant. Up to 76 evaluable participants will be accrued across the 3 stages.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Body weight 40-100 kg.
3. Capable of swallowing oral medication.
4. The Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Life expectancy >3 months.
6. Histologically or cytologically confirmed diagnosis of a solid tumor. Note: Participants with lymphomas may be enrolled. Participants with leukemia should not be included.
7. Presence of locally advanced or metastatic disease that is not amenable to surgery, radiation therapy, or chemotherapy with curative intent.
8. Cancer progression on or after standard therapy or cancer for which no standard therapy is available.
9. Discontinuation of all anticancer therapies ≥3 weeks before initiation of study treatment. Note: Prior treatment with antiangiogenic therapies (for example, bevacizumab, sunitinib, sorafenib, or investigational antiangiogenic agents) is allowed.
10. Acute toxic effects (as evaluated by CTCAE, Version 3.0) of any prior therapy resolved as shown below:

    * Neuropathy - Grade ≤2 (Stage 1 and 2)
    * Neuropathy - Grade ≤1 (Stage 3)
    * Alopecia - Grade ≤2 (all stages)
    * Fatigue - Grade ≤2 (all stages)
    * All others - Grade ≤1 (all stages)
11. Required baseline laboratory data:

    * Absolute neutrophil count ≥1,500/cubic millimeter (mm^3)
    * Platelets ≥100,000/mm^3
    * Hemoglobin ≥9.0 grams/deciliter (g/dL)
    * Serum total bilirubin <ULN; ≤1.5x ULN is acceptable if there is liver involvement secondary to tumor
    * Serum Alanine transaminase and Aspartate transaminase <ULN; ≤2.5x ULN is acceptable if there is liver involvement secondary to tumor
    * Serum alkaline phosphatase ≤2.5x ULN regardless of liver involvement with tumor
    * Serum albumin ≥3.0 g/dL
    * Serum creatinine ≤2.0 milligrams/liter (mg/L)
    * Urine protein <2+ by dipstick (or spot urinary protein: creatinine ratio <1.0 mg/dL:mg/dL, if quantitative method used)
    * Prothrombin time and Activated partial thromboplastin time ≤ULN
    * Serum beta-human chorionic gonadotropin (HCG) negative
12. Willingness, if not postmenopausal or surgically sterile, to abstain from sexual intercourse or employ an effective method of contraception during the study periods.
13. Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, and study restrictions.
14. Ability to provide written informed consent.
15. Evidence of a personally signed informed consent indicating that the participant is aware of the neoplastic nature of his or her disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential benefits, possible side effects, potential risks and discomforts, and other pertinent aspects of study participation.
16. An interval of >2 weeks from corticosteroid dose stabilization prior to obtaining the baseline MRI scan in participants with CNS malignancy.

Exclusion Criteria:

1. Unstable brain or leptomeningeal disease based on history and physical examination. Note: Enrollment of participants with central nervous system metastases is permitted if such disease is considered stable in the judgment of the investigator. A baseline magnetic resonance imaging (MRI) scan of the brain is required if there is clinical suspicion of central nervous system metastases, hemorrhage, thromboembolism, or increased intracranial pressure.
2. Any of the following in the past 3 months: myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, congestive heart failure (New York Heart Association Class III or IV), cerebrovascular accident, transient ischemic attack, any other arterial thromboembolic event, or pulmonary embolism.
3. Known coagulopathy or bleeding diathesis.
4. Known history of drug-induced liver injury.
5. Resting systolic blood pressure >180 millimeters of mercury (mmHg) or diastolic blood pressure >110 mmHg.
6. Evidence of ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infections). Note: Participants with localized fungal infections of skin or nails are eligible.
7. Pregnancy or breast-feeding.
8. Ongoing alcohol or drug addiction.
9. Prior exposure to PTC299.
10. Exposure to another investigational drug within 4 weeks prior to the study treatment.
11. Concurrent participation in another therapeutic treatment trial.
12. History of major surgical procedure within 14 days prior to enrollment in this study.
13. Psychological, social, familial, or geographical factors that would prevent regular follow up.
14. Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, ECG finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the participant; alter the absorption, distribution, metabolism or excretion of the study drug; or impair the assessment of study results.
15. History of severe hypersensitivity reactions to docetaxel or polysorbate 80. Note: This criterion applies to Stage 3 study candidates only.
16. Presence of malignancy that is refractory to docetaxel (that is, best response with prior docetaxel was progressive disease at first assessment). Note: This criterion applies to Stage 3 study candidates only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-07-03 (Actual); Primary Completion 2012-02-24 (Actual); Study Completion 2012-02-24 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of PTC299 within the tested dose range. | 6 Weeks
  To analyze the MTD of PTC299 within the tested dose range for use in further clinical trials in participants with advanced cancer.

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs) | From Baseline up to Week 246
  The relationship of TEAEs and SAEs to the study drugs will be assessed as: definite related, probable related, possible related, unlikely related, and unrelated. The severity of TEAEs will be graded using the Common Terminology Criteria for Adverse Events, Version 3.0 as: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening), or Grade 5 (fatal). A summary of serious and all other non-serious adverse events, regardless of causality, will be located in the Reported Adverse Events module.
Number of Participants With a Clinically Relevant Abnormal Clinical Laboratory Parameter | From Baseline up to Week 246
  Number of participants with an abnormal clinical laboratory parameter considered clinically relevant by the Investigator will be reported. Clinical laboratory tests will include hematology, coagulation, biochemistry, and urinalysis. A summary of serious and all other non-serious adverse events, regardless of causality, will be located in the Reported Adverse Events module.
Number of Participants With a Clinically Significant Abnormal Electrocardiogram (ECG) | From Baseline up to Week 246
  Number of participants with an abnormal ECG considered clinically significant by the Investigator will be reported. A summary of serious and all other non-serious adverse events, regardless of causality, will be located in the Reported Adverse Events module.
Number of Participants With a Dose-limiting Toxicity (DLT) | From Baseline up to Week 246
  DLT defined as occurrence of any of the following considered related to PTC299 administration:
  Stage 1
  * Other Grade ≥3 PTC299-related toxicities.
  * Failure to complete ≥80% (that is, ≥45 doses) of planned 56 doses of PTC299 treatment course due to PTC299-related toxicities.
  Stages 2, 3, 4
  * Grade ≥3 serum bilirubin (>3.0*upper limits of normal [ULN]), whether or not serum ALT or AST is elevated
  * Other Grade ≥3 PTC299-related toxicities.
  * Change in serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) from baseline (Grade 0) to Grade ≥2 (>2.5*ULN).
  Stages 1, 2, 3, 4
  * Grade ≥2 PTC299-related vomiting despite maximal oral antiemetic therapy, or requirement for intravenous antiemetics to control the nausea and vomiting.
  * Grade ≥2 proteinuria.
  * On-treatment serum ALT or AST of Grade ≥3 (>5.0*ULN).
  * Failure to recover from PTC299-related AEs to baseline AE levels by Days 42, 49, 28, and 22 of cycle for Stages 1, 2, 3, and 4, respectively.
Change From Baseline in the Circulating Concentrations of Vascular Endothelial Growth Factor (VEGF) | Baseline; Stage 1: Days 1, 14, and 28 in Cycle 1 and Days 1 and 28 of next cycles; Stage 2: Days 1, 21, and 42 in Cycle 1 and Day 42 of next cycles; Stage 3: Day 1 of each cycle; Stage 4: Days 1, 8, 15, and 22 in Cycle 1 and Day 1 of next cycles
  Two blood samples (6 milliliters [mL] of venous blood for plasma and 4 mL of venous blood for serum) are to be obtained for assessment of circulating VEGF. Participants can be evaluated for up to 14 cycles per Stage.
Proportion of Participants With a VEGF Response | Baseline; Stage 1: Days 1, 14, and 28 in Cycle 1 and Days 1 and 28 of next cycles; Stage 2: Days 1, 21, and 42 in Cycle 1 and Day 42 of next cycles; Stage 3: Day 1 of each cycle; Stage 4: Days 1, 8, 15, and 22 in Cycle 1 and Day 1 of next cycles
  VEGF-A response is defined as ≥25% decrease relative to the baseline concentration at any time during study treatment. Two blood samples (6 mL of venous blood for plasma and 4 mL of venous blood for serum) are to be obtained for assessment of circulating VEGF. Participants can be evaluated for up to 14 cycles per Stage.
Change From Baseline in Ktrans | Baseline; Stage 1: Day 3 and Day 26 of Cycle 1; Stage 2: Day 42 of Cycle 1
  Ktrans defined as volume transfer constant between blood plasma and extra-cellular extra-vascular space.
Area Under the Concentration Blood Normalized, 90 Seconds (AUCBN90) in a Target Tumor Lesion | Baseline; Stage 1: Day 3 and Day 26 of Cycle 1; Stage 2: Day 42 of Cycle 1
  AUCBN90 defined as blood-normalized area under the tumor enhancement curve over the first 90 seconds post-injection.
Tumor Metabolism as Assessed by Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) | Every 6 weeks per cycle in Stages 1, 2, 3, and 4 (each stage could include up to 14 cycles)
  Change in tumor metabolism as assessed by changes in FDG-PET standardized uptake value (SUV) in a target tumor lesion.
Change From Baseline in Tumor Size | Every 6 weeks per cycle in Stages 1, 2, 3, and 4 (each stage could include up to 14 cycles)
  The change in tumor size from baseline is to be described by dose at each assessment and the greatest change during the study will be computed.
Proportion of Participants With an On-treatment Tumor Response | Every 6 weeks per cycle in Stages 1, 2, 3, and 4 (each stage could include up to 14 cycles)
  Tumor response defined by Response Evaluation Criteria in Solid Tumors (RECIST). Definitions of tumor lesion responses: Complete response (CR) - disappearance of all target lesions; Partial response (PR) - ≥30% decrease in the sum of the longest dimensions of the target lesions, taking as a reference the baseline sum of the longest dimensions; Progressive disease (PD) - ≥20% increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of 1 or more new lesions; Stable disease (SD) - neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD, taking as a reference the smallest sum of the longest dimensions since the treatment started.
Change From Baseline in Tumor Marker Response | Every 6 weeks per cycle in Stages 1, 2, 3, and 4 (each stage could include up to 14 cycles)
  Tumor marker response defined as a reduction by ≥50% in the tumor marker value relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Schwartz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: PTC Therapeutics, Inc. Webpage — http://www.ptcbio.com